CLINICAL TRIAL: NCT00072436
Title: A Phase I Trial of Gemcitabine Followed by a Short Infusion of Flavopiridol in Patients With Solid Tumors
Brief Title: Gemcitabine Hydrochloride and Alvocidib in Treating Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00038; 6051; P30CA006516 (NIH); U01CA062490 (NIH); CDR0000339727 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2003-11-04; First posted 2003-11-06 (Estimated); Last update posted 2013-07-02 (Estimated); Status verified 2013-07

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — Gemcitabine; alvocidib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Some patients receive an initial dose of alvocidib IV over 1-7 hours on day 1 (course 0). Beginning 1 week later and for all subsequent courses, all patients receive gemcitabine hydrochloride IV over 60-150 minutes on days 1 and 15 and alvocidib IV over 1-7 hours on days 2 and 16. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3-6 patients receive escalating doses of gemcitabine hydrochloride and alvocidib until the MTD is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, up to 10 additional patients receive treatment at that dose.
  Interventions: Drug: gemcitabine hydrochloride; Drug: alvocidib; Other: pharmacological study

INTERVENTIONS:
Drug: gemcitabine hydrochloride — Given IV
  Other Names: dFdC; difluorodeoxycytidine hydrochloride; gemcitabine; Gemzar
Drug: alvocidib — Given IV
  Other Names: FLAVO; flavopiridol; HMR 1275; L-868275
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This phase I trial is studying the side effects and best dose of gemcitabine hydrochloride and alvocidib in treating patients with solid tumors. Drugs used in chemotherapy, such as gemcitabine hydrochloride and alvocidib, use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose of gemcitabine and flavopiridol in patients with solid tumors.

SECONDARY OBJECTIVES:

I. Determine the safety profile and toxic effects of this regimen in these patients.

II. Determine the pharmacokinetics of flavopiridol with and without gemcitabine in these patients.

III. Determine, using pharmacodynamic assays, the activity of flavopiridol as a cdk inhibitor in these patients.

IV. Determine, using pharmacodynamic assays, the markers of this regimen in these patients.

OUTLINE: This is a dose-escalation, multicenter study.

Some patients receive an initial dose of alvocidib IV over 1-7 hours on day 1 (course 0). Beginning 1 week later and for all subsequent courses, all patients receive gemcitabine hydrochloride IV over 60-150 minutes on days 1 and 15 and alvocidib IV over 1-7 hours on days 2 and 16. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of gemcitabine hydrochloride and alvocidib until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, up to 10 additional patients receive treatment at that dose.

Patients are followed at 30 days after study completion.

ELIGIBILITY:
Inclusion Criteria:

* Negative pregnancy test
* Fertile patients must use effective contraception
* No active infection
* No severe malnutrition
* No more than 2 prior chemotherapy regimens:

  * Prior combined modality therapy (e.g., full-dose chemotherapy with radiosensitizing chemotherapy and radiotherapy) is considered 1 prior regimen if all therapy was delivered as part of 1 comprehensive treatment plan
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* No other concurrent chemotherapy
* At least 6 months since prior radiotherapy to the lung parenchyma or mediastinum and no evidence of radiation pneumonitis on chest CT scan
* At least 4 weeks since other prior radiotherapy and recovered
* No prior radiotherapy to more than 50% of marrow volume
* No concurrent radiotherapy
* Histologically confirmed solid tumor for which gemcitabine is a treatment option OR for which no efficacious therapy exists
* Must meet criteria for 1 of the following:

  * Measurable disease:

    * At least 1 unidimensionally measurable lesion at least 20 mm by conventional techniques OR at least 10 mm by spiral CT scan
  * Nonmeasurable disease, including any of the following:

    * Small lesions (less than 20 mm by conventional techniques OR less than 10 mm by spiral CT scan)
    * Bone lesions
    * Cytologically positive pleural or peritoneal disease
    * Elevated tumor markers (e.g., carcinoembryonic antigen, CA 125, CA 19-9, or other tumor marker)
    * Multinodular or confluent nonmeasurable pulmonary, hepatic, adrenal, intra-abdominal, or skin metastases
    * No active CNS metastases
    * Previously treated CNS metastases must be stable with no symptoms for 4 weeks after completion of treatment AND patient must be off steroid therapy or on a stable dose for at least the past 2 weeks
    * No known leptomeningeal metastases
* Performance status:

  * ECOG 0-1
* Hematopoietic:

  * Absolute neutrophil count at least 1,500/mm3;
  * Platelet count at least 100,000/mm3
* Hepatic:

  * Bilirubin no greater than 1.5 mg/dL;
  * SGOT no greater than 2.5 times upper limit of normal
* Renal:

  * Creatinine no greater than 1.5 mg/dL OR
  * Creatinine clearance at least 50 mL/min
* Cardiovascular:

  * None of the following within the past 6 months:

    * Myocardial infarction;
    * Unstable angina;
    * Transient ischemic attack;
    * Cerebrovascular accident

      * No new cardiac arrhythmia possibly related to cardiac ischemia;
      * No large and potentially symptomatic pericardial effusion;
      * No cardiac disease that would preclude study participation
* Pulmonary:

  * No pulmonary embolism within the past 6 months;
  * No large and potentially symptomatic pleural effusion;
  * No pulmonary disease that would preclude study participation
* Gastrointestinal:

  * No intractable emesis;
  * No grade 2 or greater chronic diarrheal disease within the past 6 months
* Not pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2003-09; Primary Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) graded by National Cancer Institute (NCI) Common Toxicity Criteria | 28 days
Maximum tolerated dose, defined as one dose level below the dose that induces DLT in more than 1/6 patients | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Shapiro, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York